CLINICAL TRIAL: NCT00557986
Title: The Effect of Primary Surgical Treatment on Survival in Patients With Metastatic Breast Cancer at Diagnosis
Brief Title: Local Surgery for Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federation of Breast Diseases Societies (Other)
Collaborators: Istanbul University (Other); Abant Izzet Baysal University (Other); Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MF07-01
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: 1-Metastatic breast cancer; 2-Surgery; 3-Survival
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (No Intervention): Standard Systemic Therapy only group (no primary surgery)
- B (Other): Surgery group
  Interventions: Procedure: Primary surgery

INTERVENTIONS:
Procedure: Primary surgery — Primary breast surgery before systemic therapy
  Arms: B

SUMMARY:
Primary treatments for metastatic breast cancer are chemotherapy and radiation therapy, and surgery is reserved for tumor related complications such as bleeding. Retrospective studies showed that surgical removal of the primary tumor improves survival of patients with metastatic breast cancer at diagnosis. We hypothesis and testing that surgical removal of the primary tumor will lead to an improvement of overall survival

DETAILED DESCRIPTION:
This is a randomised, controled clinical trial. Our aim is to observe whether primary surgery improves survival in metastatic breast cancer. Women who have metastatic breast cancer at the initial diagnosis will be included in the study. There will be two study arms: primary surgery and systemic chemotherapy groups.

In the primary surgery group patients will have adjuvant therapies after they had the proper surgery. In the systemic chemotherapy group patients will be followed after their initial therapy and will have surgery only if they have locoregional problems (such as wide necrosis or bleeding, etc). During the follow-up period, patients will be seen in every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women with metastatic breast cancer at the initial diagnosis

Exclusion Criteria:

* Women needs breast surgery at the time of initial diagnosis (such as bleeding, necrosis, etc)
* who have systemic morbidity that do not allows her to be in the trial,
* who have synchronous breast cancer at the contralateral breast,
* who have a previous cancer history or another primary cancer history and metastasis at the past,
* who have palpable lymph node/nodes at the contralateral axilla,
* who do not agree to participate the trial

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2007-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Measure: all cause mortality | 5 years

SECONDARY OUTCOMES:
Quality of life | 5 year
mordities | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Atilla Soran, MD, MPH, Study Chair — University of Pittsburgh; Atilla Soran, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (7):
- Turkey (Türkiye) (7):
  - Cukurova University, Adana
  - Ankara Onkoloji Hastanesi, Ankara
  - Adnan Menderes University, Aydin
  - Izzet Baysal University, Bolu
  - Istanbul University Medical faculty, Istanbul
  - Marmara Univesity School of Medicine, Istanbul
  - Cumhuriyet University Medical School, Sivas

REFERENCES:
- [Background] Rapiti E, Verkooijen HM, Vlastos G, Fioretta G, Neyroud-Caspar I, Sappino AP, Chappuis PO, Bouchardy C. Complete excision of primary breast tumor improves survival of patients with metastatic breast cancer at diagnosis. J Clin Oncol. 2006 Jun 20;24(18):2743-9. doi: 10.1200/JCO.2005.04.2226. Epub 2006 May 15. PMID 16702580
- [Background] Babiera GV, Rao R, Feng L, Meric-Bernstam F, Kuerer HM, Singletary SE, Hunt KK, Ross MI, Gwyn KM, Feig BW, Ames FC, Hortobagyi GN. Effect of primary tumor extirpation in breast cancer patients who present with stage IV disease and an intact primary tumor. Ann Surg Oncol. 2006 Jun;13(6):776-82. doi: 10.1245/ASO.2006.03.033. Epub 2006 Apr 17. PMID 16614878
- [Derived] Soran A, Ozmen V, Ozbas S, Karanlik H, Muslumanoglu M, Igci A, Canturk NZ, Utkan Z, Evrensel T, Sezgin E; MF07-01 Study Group. Primary Surgery with Systemic Therapy in Patients with de Novo Stage IV Breast Cancer: 10-year Follow-up; Protocol MF07-01 Randomized Clinical Trial. J Am Coll Surg. 2021 Dec;233(6):742-751.e5. doi: 10.1016/j.jamcollsurg.2021.08.686. Epub 2021 Sep 13. PMID 34530124
- [Derived] Soran A, Soyder A, Ozbas S, Ozmen V, Karanlik H, Igci A, Muslumanoglu M, Evrensel T, Canturk Z, Utkan Z, Ozaslan C, Uras C, Ugurlu U, Col C, Cabioglu N, Uzunkoy A, Gulluoglu BM, Erdem E, Konca C, Sezgin E; Breast Health Working Group International (supported by the Turkish Federation of Breast Disease Societies). The role of loco-regional treatment in long-term quality of life in de novo stage IV breast cancer patients: protocol MF07-01Q. Support Care Cancer. 2021 Jul;29(7):3823-3830. doi: 10.1007/s00520-020-05905-z. Epub 2020 Nov 26. PMID 33242163
- [Derived] Soran A, Ozmen V, Ozbas S, Karanlik H, Muslumanoglu M, Igci A, Canturk Z, Utkan Z, Ozaslan C, Evrensel T, Uras C, Aksaz E, Soyder A, Ugurlu U, Col C, Cabioglu N, Bozkurt B, Uzunkoy A, Koksal N, Gulluoglu BM, Unal B, Atalay C, Yildirim E, Erdem E, Salimoglu S, Sezer A, Koyuncu A, Gurleyik G, Alagol H, Ulufi N, Berberoglu U, Dulger M, Cengiz O, Sezgin E, Johnson R. Randomized Trial Comparing Resection of Primary Tumor with No Surgery in Stage IV Breast Cancer at Presentation: Protocol MF07-01. Ann Surg Oncol. 2018 Oct;25(11):3141-3149. doi: 10.1245/s10434-018-6494-6. Epub 2018 May 17. PMID 29777404
- [Derived] Soran A, Ozbas S, Kelsey SF, Gulluoglu BM. Randomized trial comparing locoregional resection of primary tumor with no surgery in stage IV breast cancer at the presentation (Protocol MF07-01): a study of Turkish Federation of the National Societies for Breast Diseases. Breast J. 2009 Jul-Aug;15(4):399-403. doi: 10.1111/j.1524-4741.2009.00744.x. Epub 2009 May 22. PMID 19496782